CLINICAL TRIAL: NCT00709111
Title: A Pilot Trial of Maraviroc for Treatment of Subjects on Antiretroviral Therapy With Suboptimal CD4 T-cell Count Recovery Despite Sustained Virologic Suppression
Brief Title: Adding Maraviroc to Antiretroviral Therapy for Suboptimal CD4 T-Cell Recovery Despite Sustained Virologic Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5256; 1U01AI068636 (NIH)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
Keywords: CCR5 antagonist; CD4 T-cell count; immune activation; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maraviroc (Experimental): Maraviroc (MVC) was taken for 24 weeks, in addition to the subject's current antiretroviral therapy (ART) drug regimen. At week 24, subjects discontinued MVC and were followed for an additional 24 weeks off MVC, but still on current ART drug regimen.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — The maraviroc doses were 150 mg orally twice daily, 300 mg orally twice daily, or 600 mg orally twice daily, depending on the pharmacokinetic interaction with a subject's pre-study ART and non-ART drug regimen according to the package insert.
  Other Names: MVC; Selzentry

SUMMARY:
Despite viral suppression, antiretroviral therapy (ART) does not restore CD4+ T-cell counts in some subjects. The purpose of this study is to assess whether adding maraviroc (MVC) to a suppressive ART will result in a significant CD4+ T-cell count increase over 24 weeks in subjects with suboptimal CD4+ T-cell recovery despite sustained virologic suppression.

DETAILED DESCRIPTION:
The majority of HIV-infected subjects with virologic suppression on antiretroviral therapy (ART) have a marked increase in CD4+ T-cell counts over the first year on treatment. However, a portion of these individuals show a suboptimal immune response and remain at an elevated risk for disease progression. The use of the CCR5 inhibitor maraviroc (MVC) is associated with enhanced CD4+ T-cell recovery in subjects who initiate ART. AIDS Clinical Trials Group (ACTG) A5256 studied the effect of ART intensification with MVC on CD4+ T-cell counts in subjects with suboptimal CD4 recovery despite sustained virologic suppression. Eligible subjects added MVC to their ART regimen, and continued MVC for 24 weeks. At week 24, subjects discontinued MVC and were followed for an additional 24 weeks off MVC.

Subjects were seen through week 48 for clinical and laboratory evaluations, including plasma HIV-1 RNA, CD4+ T-cell count, and safety laboratories. Subjects had 2 baseline visits prior to starting MVC. Study visits were scheduled at weeks 4, 8, 12, 16, 22, 24, 36, 46, and 48. CD4+ T-cell counts were measured at every study visit and HIV-1 RNA at weeks 12, 24, 36, and 48, regardless of treatment status. Measures of activation, T-cell maturation, and apoptosis were performed at all weeks except 4, 8, and 16. At the end of the study, the pre-entry, entry, week 12, 22, 24, and 36 samples for the HIV-1 RNA by single-copy assay (SCA) were run. The week 46 and 48 samples were not run.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* On ART for at least 48 weeks prior to study entry with a regimen that includes three or more antiretroviral medications
* No change in ART regimen for at least 24 weeks prior to study entry
* Screening CD4+ T-cell count less than 250 obtained within 60 days prior to study entry
* Stable CD4+ T-cell count for at least 48 weeks prior to study entry (as assessed by an estimated CD4+ T-cell count slope between -20 and +20 cells/year)
* Screening HIV-1 RNA below the limit of detection using an FDA-approved assay obtained within 60 days prior to study entry
* All other plasma HIV-1 RNA measurements in the 48 weeks prior to study entry must be below the limit of detection
* Laboratory values obtained within 60 days prior to study entry:

  * Absolute neutrophil count (ANC) >=750/µL
  * Hemoglobin >=9.0 g/dL for female subjects and >=10.0 g/dL for male subjects
  * Platelet count >=50,000/ µL
  * Calculated creatinine clearance (CrCl) >=30 mL/min
  * Aspartate aminotransferase (serum glutamic oxaloacetic transaminase), alanine aminotransferase (serum glutamic pyruvic transaminase), and alkaline phosphatase <=5 X Upper Limit of Normal (ULN)
  * Direct bilirubin <=2.5 X ULN
* Females of reproductive potential will need a negative serum or urine pregnancy test within 48 hours prior to study entry
* Agree not to participate in the conception process, and if participating in sexual activity that could lead to pregnancy, the subject/partner must use at least two reliable forms of contraceptives while receiving study treatment and for 6 weeks after stopping study treatment.

Exclusion Criteria:

* Unstable clinical condition
* Currently breast-feeding or pregnant
* Use of immunomodulators or cancer chemotherapy or radiation treatment within 12 months prior to study entry
* An acute AIDS-defining illness within 60 days prior to study entry
* Known allergy/sensitivity or hypersensitivity to components of MVC, including allergy or hypersensitivity to soya lecithin, soya or peanuts
* Active drug or alcohol abuse that, in the opinion of the investigator, would interfere with adherence to study regimens
* Serious illness requiring systemic treatment and/or hospitalization within 60 days prior to study entry
* Receipt of a vaccine within 30 days prior to study entry
* Current or previous use of a CCR5 inhibitor
* Plan to change background ART regimen within 24 weeks after study entry
* Receipt of experimental or non-experimental medications for the purpose of raising CD4+ T-cell counts within 6 months prior to study entry

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Wilkin, MD, MPH, Study Chair — Cornell Clinical Research Site; Roy Gulick, MD, MPH, Study Chair — Cornell HIV Clinical Trials Unit
Locations (29):
- United States (29):
  - Alabama Therapeutics CRS (5801), Birmingham, Alabama
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Stanford CRS (501), Palo Alto, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - Ucsf Aids Crs (801), San Francisco, California
  - Georgetown University CRS (GU CRS) (1008), Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS (901), Miami, Florida
  - The Ponce de Leon Ctr. CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - IHV Baltimore Treatment CRS (4651), Baltimore, Maryland
  - Johns Hopkins Adult AIDS CRS (201), Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Boston Medical Center ACTG CRS (104), Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - Cornell CRS (7804), New York, New York
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - AIDS Care CRS (1108), Rochester, New York
  - Univ. of Rochester ACTG CRS (1101), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS (1601), Durham, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - MetroHealth CRS (2503), Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS (2301), Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - Pittsburgh CRS (1001), Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Peabody Health Ctr. CRS (31443), Dallas, Texas
  - Houston AIDS Research Team CRS (31473), Houston, Texas

REFERENCES:
- [Background] Fadel H, Temesgen Z. Maraviroc. Drugs Today (Barc). 2007 Nov;43(11):749-58. doi: 10.1358/dot.2007.43.11.1131763. PMID 18174962
- [Background] MacArthur RD, Novak RM. Reviews of anti-infective agents: maraviroc: the first of a new class of antiretroviral agents. Clin Infect Dis. 2008 Jul 15;47(2):236-41. doi: 10.1086/589289. PMID 18532888
- [Result] Wilkin T, Lalama C, Tenorio A, Landay A, Ribaudo H, McKinnon J, Gandhi R, Mellors J, Currier J, and Gulick R. Maraviroc Intensification for Suboptimal CD4+ Cell Response Despite Sustained Virologic Suppression: ACTG 5256. 17th Conference on Retroviruses and Opportunistic Infections, San Francisco, CA, February 16-19, 2010.
- [Result] Wilkin T, Lalama C, Tenorio A, Landay A, Fox L, McKinnon J, Gandhi R, Mellors J, Currier J, Gulick R. ACTG 5256: Effect of adding and removing maraviroc (MVC) on immune activation in participants on suppressive antiretroviral therapy (ART). 18th Conference on Retroviruses and Opportunistic Infections, Boston, MA, February 27-March 02, 2011.
- [Result] Hilldorfer B, Lalama C, McKinnon J, Coombs B, Tenorio A, Fox L, Gandhi R, Ribaudo H, Currier J, Gulick R, Wilkin TJ, Mellors J. Effects of Maraviroc (MVC) on Residual Low-Level Viremia in Patients on Suppressive Antiretroviral Therapy (ART): Results from ACTG 5256. 6th IAS Conference on HIV Pathogenesis, Treatment and Prevention, Rome, Italy, July 17-20, 2011.
- [Derived] Wilkin TJ, Lalama CM, McKinnon J, Gandhi RT, Lin N, Landay A, Ribaudo H, Fox L, Currier JS, Mellors JW, Gulick R, Tenorio AR. A pilot trial of adding maraviroc to suppressive antiretroviral therapy for suboptimal CD4(+) T-cell recovery despite sustained virologic suppression: ACTG A5256. J Infect Dis. 2012 Aug 15;206(4):534-42. doi: 10.1093/infdis/jis376. Epub 2012 Jun 27. PMID 22740718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at 29 AIDS Clinical Trials Units in the United States between January 14, 2009 and May 4, 2009
Pre-assignment Details: 34 enrolled
Period: Overall Study
Arm/Group | Maraviroc
Started | 34
Week 22/24 | 33
Completed | 32
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Unable to attend clinic visits | 1

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc
Number analyzed (Participants) | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [47 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 32
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 24
  Black Non-Hispanic | 6
  Hispanic (Regardless of Race) | 4
Baseline CD4+ T-cell count [Median (Inter-Quartile Range); unit: cells/mm^3] — Baseline CD4+ T-cell count is the average (mean) of the pre-entry and entry values
  cells/mm^3 | 153 [119 to 203]
Baseline CD4 percentage [Median (Inter-Quartile Range); unit: % of total lymphocytes] — Baseline CD4 percentage is the average (mean) of the pre-entry and entry values
  % of total lymphocytes | 13 [10 to 17]
Baseline CD8+ T-cell count [Median (Inter-Quartile Range); unit: cells/mm^3] — Baseline CD8+ T-cell count is the average (mean) of the pre-entry and entry values
  cells/mm^3 | 559 [416 to 872]
Time with suppressed HIV-1 RNA prior to study entry [Median (Inter-Quartile Range); unit: years] — Four (4) participants had no documentation or recall of the date when they became suppressed (HIV-1 RNA <400 copies/ml)
  years | 3.0 [1.8 to 4.5]

OUTCOME MEASURES:

1. Primary Outcome: Change in CD4+ T-cell Count
Description: Change was calculated as the week 24 CD4+ T-cell count (average of the week 22 and week 24 values) minus the baseline CD4+ T-cell count (average of pre-entry and entry values).
Time Frame: From baseline to week 24
Population: As-treated: Only participants with either a week 22 CD4+ T-cell count or a week 24 CD4+ T-cell count obtained while receiving MVC without change in background regimen were included.
Measure: Median (90% Confidence Interval); unit: cells/mm^3
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
cells/mm^3 | 12 [1 to 22]
Statistical Analysis 1: Comparison: Maraviroc; The change in CD4+ T-cell count from baseline to week 24 was compared against the null hypothesis of change <20 cells/mm^3. The study was powered to yield 80% power to show that there was >=20 cells/mm^3 increase in CD4+ T-cell count assuming an underlying change in CD4+ T-cell counts induced by MVC of 50 cells/mm^3, a standard deviation of 60 cells/mm^3 around the mean CD4+ T-cell count change, 10% lost-to-follow-up or premature MVC discontinuation rate, and one-sided type 1 error of 0.05; Test type: Superiority or Other; p = 0.97, Wilcoxon signed-rank, 1-sided — The p-value is one-sided with a nominal level of 0.05

2. Secondary Outcome: Proportion of Participants Achieving a 50-cell Increase in CD4+ T-cell Count
Description: Baseline was defined as the average of pre-entry and entry values. Week 24 was defined as the average of the week 22 and week 24 values.
Time Frame: From baseline to week 24
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
proportion of participants | 0.06 [0.01 to 0.18]

3. Secondary Outcome: Within-subject CD4+ T-cell Count Slopes
Description: The estimated mean slope was summarized across the population by using generalized estimating equations. Baseline was defined as the average of pre-entry and entry values. Week 24 was defined as the average of the week 22 and week 24 values.
Time Frame: From baseline through week 24
Population: As-treated: Participants with CD4+ T-cell counts available at least through visit week 22 while receiving MVC without change in background regimen were included.
Measure: Mean (90% Confidence Interval); unit: cells/mm^3/year
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
cells/mm^3/year | 24.7 [2.9 to 46.4]

4. Secondary Outcome: Change From Within-subject Pre-treatment CD4+ T-cell Count Slopes to Corresponding Within-subject CD4+ T-cell Count Slopes From Baseline Through Week 24
Description: The estimated mean change in slopes was summarized across the population by using generalized estimating equations. Pre-treatment CD4+ T-cell counts (from at least 48 weeks prior to study entry) were recorded at screening from patient source documentation. Baseline was defined as the average of pre-entry and entry values. Week 24 was defined as the average of the week 22 and week 24 values.
Time Frame: From pre-treatment through week 24
Population: as for outcome 3
Measure: Mean (90% Confidence Interval); unit: cells/mm^3/year
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
cells/mm^3/year | 25.2 [2.1 to 48.3]

5. Secondary Outcome: Change in CD4+ T-cell Count
Description: Change was calculated as week 36 CD4+ T-cell count minus the week 24 CD4+ T-cell count (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 36
Population: As-treated: Only participants that were included in the primary week 24 analysis, i.e. change from baseline to week 24, and with a week 36 CD4+ T-cell count obtained while receiving background regimen were included.
Measure: Median (90% Confidence Interval); unit: cells/mm^3
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
cells/mm^3 | -3 [-16 to 7]

6. Secondary Outcome: Change in CD4+ T-cell Count
Description: Change was calculated as week 48 CD4+ T-cell count (average of week 46 and week 48) minus the week 24 CD4+ T-cell count (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 48
Population: As-treated: Only participants that were included in the primary week 24 analysis, i.e. change from baseline to week 24, and with either a week 46 CD4+ T-cell count or a week 48 CD4+ T-cell count obtained while receiving background regimen were included.
Measure: Median (90% Confidence Interval); unit: cells/mm^3
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
cells/mm^3 | 7 [-5 to 18]

7. Secondary Outcome: Change in CD4 Percentage
Description: Change was calculated as the week 24 CD4 percentage (average of the week 22 and week 24 values) minus the baseline CD4 percentage (average of pre-entry and entry values).
Time Frame: From baseline to week 24
Population: As-treated: Only participants with either a week 22 CD4 percentage or a week 24 CD4 percentage obtained while receiving MVC without change in background regimen were included.
Measure: Median (90% Confidence Interval); unit: % of total lymphocytes
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
% of total lymphocytes | 0.5 [0 to 0.9]

8. Secondary Outcome: Within-subject CD4 Percentage Slopes
Description: as for outcome 3
Time Frame: From baseline through week 24
Population: As-treated: Participants with CD4 percentage available at least through visit week 22 while receiving MVC without change in background regimen were included. Four of these subjects did not have pre-treatment (from at least 48 weeks prior to study entry) CD4 percentage results available.
Measure: Mean (90% Confidence Interval); unit: % of total lymphocytes/year
Arm/Group | Maraviroc
Number analyzed (Participants) | 28
% of total lymphocytes/year | -0.3 [-2.2 to 1.6]

9. Secondary Outcome: Change From Within-subject Pre-treatment CD4 Percentage Slopes to Corresponding Within-subject CD4 Percentage Slopes From Baseline Through Week 24
Description: The estimated mean change in slopes was summarized across the population by using generalized estimating equations. Pre-treatment CD4 percentage (from at least 48 weeks prior to study entry) were recorded at screening from patient source documentation. Baseline was defined as the average of pre-entry and entry values. Week 24 was defined as the average of the week 22 and week 24 values.
Time Frame: From pre-treatment through week 24
Population: as for outcome 8
Measure: Mean (90% Confidence Interval); unit: % of total lymphocytes/year
Arm/Group | Maraviroc
Number analyzed (Participants) | 28
% of total lymphocytes/year | -1.0 [-3.0 to 1.1]

10. Secondary Outcome: Change in CD4 Percentage
Description: Change was calculated as week 36 CD4 percentage minus the week 24 CD4 percentage (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 36
Population: As-treated: Only participants that were included in the primary week 24 analysis, i.e. change from baseline to week 24, and with a week 36 CD4 percentage obtained while receiving background regimen were included.
Measure: Median (90% Confidence Interval); unit: % of total lymphocytes
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
% of total lymphocytes | 0.2 [-0.1 to 1.0]

11. Secondary Outcome: Change in CD4 Percentage
Description: Change was calculated as week 48 CD4 percentage (average of week 46 and week 48) minus the week 24 CD4 percentage (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 48
Population: As-treated: Only participants that were included in the primary week 24 analysis, i.e. change from baseline to week 24, and with either a week 46 CD4 percentage or a week 48 CD4 percentage obtained while receiving background regimen were included.
Measure: Median (90% Confidence Interval); unit: % of total lymphocytes
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
% of total lymphocytes | 0.5 [0 to 1.5]

12. Secondary Outcome: Number of Subjects Who Experience a Grade 2, 3 or 4 Signs and Symptoms, Grade 3 or 4 Laboratory Abnormalities, or Death.
Description: Events with date of onset or specimen date prior to first dose of MVC or after the last dose of MVC were excluded. Signs and symptoms with a date of onset the same as the first dose of MVC were excluded if confirmed by the site to be before the first dose. Lab abnormalities with the date of specimen the same as the date of the first dose of MVC were excluded on the assumption that the specimen was drawn before the first dose. Grading used the Division of AIDS (DAIDS) 2004 Severity of Adverse Events Tables, where Grade 1=Mild, 2=Moderate, 3=Severe, 4=Potentially life-threatening.
Time Frame: From baseline through week 24
Population: As-treated: Participants who initiated treatment were included. Follow-up while receiving MVC without change in background regimen were included.
Measure: Number; unit: participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 34
participants
  grade>=2 signs/symptoms or grade>=3 lab abnorm. | 15
  deaths | 0

13. Secondary Outcome: Change in Percentage of CD4+ T-cells That Are: naïve (%CD45RA+CCR7+), Central Memory (%CD45RA-CCR7+), Effector Memory (%CD45RA-CCR7-), Effector (%CD45RA+CCR7-), %HLA-DR+CD38+, %CD38+, %Ki67+, %caspase3+, %Bcl-2-, and %CD57+
Description: Change was calculated as the week 24 result (average of the week 22 and week 24 values) minus the baseline result (average of pre-entry and entry values).
Time Frame: From baseline to week 24
Population: As-treated: Only participants with either a week 22 result or a week 24 result obtained while receiving MVC without change in background regimen were included.
Measure: Median (90% Confidence Interval); unit: % of CD4+ T-cells
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
% of CD4+ T-cells
  naïve (%CD45RA+CCR7+) | -1.3 [-3.0 to 0.3]
  central memory (%CD45RA-CCR7+) | -4.8 [-7.9 to -1.9]
  effector memory (%CD45RA-CCR7-) | 5.8 [2.5 to 10.6]
  effector (%CD45RA+CCR7-) | 0.7 [0 to 0.9]
  %HLA-DR+CD38+ | -1.3 [-1.8 to -0.3]
  %CD38+ | -14.8 [-19.6 to -9.3]
  %Ki67+ | -1.0 [-1.5 to -0.5]
  %caspase3+ | -1.1 [-1.4 to -0.6]
  %Bcl-2- | 0.7 [0 to 1.3]
  %CD57+ | 1.8 [1.0 to 2.7]

14. Secondary Outcome: Change in Percentage of CD8+ T-cells That Are: naïve (%CD45RA+CCR7+), Central Memory (%CD45RA-CCR7+), Effector Memory (%CD45RA-CCR7-), Effector (%CD45RA+CCR7-), %HLA-DR+CD38+, %CD38+, %Ki67+, %caspase3+, %Bcl-2-, and %CD57+
Description: as for outcome 13
Time Frame: From baseline to week 24
Population: as for outcome 13
Measure: Median (90% Confidence Interval); unit: % of CD8+ T-cells
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
% of CD8+ T-cells
  naïve (%CD45RA+CCR7+) | -3.3 [-5.4 to -1.7]
  central memory (%CD45RA-CCR7+) | -1.0 [-1.9 to -0.5]
  effector memory (%CD45RA-CCR7-) | 2.5 [0.8 to 6.0]
  effector (%CD45RA+CCR7-) | 2.0 [0.2 to 6.6]
  %HLA-DR+CD38+ | -1.4 [-3.0 to -0.3]
  %CD38+ | -14.2 [-19.5 to -8.7]
  %Ki67+ | -0.1 [-0.3 to 0.1]
  %caspase3+ | -0.7 [-0.9 to -0.4]
  %Bcl-2- | 0.5 [-0.1 to 0.8]
  %CD57+ | 3.6 [1.0 to 5.6]

15. Secondary Outcome: Change in Percentage of CD4+ T-cells That Are: naïve (%CD45RA+CCR7+), Central Memory (%CD45RA-CCR7+), Effector Memory (%CD45RA-CCR7-), Effector (%CD45RA+CCR7-), %HLA-DR+CD38+, %CD38+, %Ki67+, %caspase3+, %Bcl-2-, and %CD57+
Description: Change was calculated as week 36 result minus the week 24 result (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 36
Population: As-treated: Only participants that were included in the primary week 24 analysis, i.e. change from baseline to week 24, and with a week 36 result obtained while receiving background regimen were included.
Measure: Median (90% Confidence Interval); unit: % of CD4+ T-cells
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
% of CD4+ T-cells
  naïve (%CD45RA+CCR7+) | 3.5 [1.1 to 5.9]
  central memory (%CD45RA-CCR7+) | -1.4 [-3.0 to -0.2]
  effector memory (%CD45RA-CCR7-) | -3.7 [-6.0 to -0.7]
  effector (%CD45RA+CCR7-) | 0.1 [-0.3 to 0.8]
  %HLA-DR+CD38+ | -0.2 [-0.5 to 0.1]
  %CD38+ | 2.8 [0.2 to 3.6]
  %Ki67+ | 0.1 [-0.2 to 0.5]
  %caspase3+ | 0.3 [0.1 to 0.4]
  %Bcl-2- | -0.6 [-0.9 to -0.2]
  %CD57+ | -0.9 [-1.7 to -0.5]

16. Secondary Outcome: Change in Percentage of CD8+ T-cells That Are: naïve (%CD45RA+CCR7+), Central Memory (%CD45RA-CCR7+), Effector Memory (%CD45RA-CCR7-), Effector (%CD45RA+CCR7-), %HLA-DR+CD38+, %CD38+, %Ki67+, %caspase3+, %Bcl-2-, and %CD57+
Description: Change was calculated as week 36 result minus the week 24 result (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 36
Population: as for outcome 15
Measure: Median (90% Confidence Interval); unit: % of CD8+ T-cells
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
% of CD8+ T-cells
  naïve (%CD45RA+CCR7+) | 2.4 [0.6 to 3.8]
  central memory (%CD45RA-CCR7+) | -0.3 [-0.9 to 0]
  effector memory (%CD45RA-CCR7-) | -5.1 [-6.7 to -3.5]
  effector (%CD45RA+CCR7-) | 2.4 [0.7 to 4.7]
  %HLA-DR+CD38+ | -0.8 [-2.0 to -0.1]
  %CD38+ | -1.6 [-5.2 to 3.3]
  %Ki67+ | 0.1 [-0.2 to 0.2]
  %caspase3+ | 0.2 [0.1 to 0.3]
  %Bcl-2- | -0.3 [-0.5 to 0.3]
  %CD57+ | -2.8 [-3.3 to -0.9]

17. Secondary Outcome: Change in Percentage of CD4+ T-cells That Are: naïve (%CD45RA+CCR7+), Central Memory (%CD45RA-CCR7+), Effector Memory (%CD45RA-CCR7-), Effector (%CD45RA+CCR7-), %HLA-DR+CD38+, %CD38+, %Ki67+, %caspase3+, %Bcl-2-, and %CD57+
Description: Change was calculated as week 48 result (average of week 46 and week 48) minus the week 24 result (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 48
Population: As-treated: Only participants that were included in the primary week 24 analysis, i.e. change from baseline to week 24, and with either a week 46 result or a week 48 result obtained while receiving background regimen were included.
Measure: Median (90% Confidence Interval); unit: % of CD4+ T-cells
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
% of CD4+ T-cells
  naïve (%CD45RA+CCR7+) | 2.1 [1.1 to 3.8]
  central memory (%CD45RA-CCR7+) | -3.1 [-6.8 to -2.0]
  effector memory (%CD45RA-CCR7-) | 0.4 [-3.0 to 2.2]
  effector (%CD45RA+CCR7-) | 1.2 [0.7 to 1.9]
  %HLA-DR+CD38+ | 0.4 [0.1 to 0.6]
  %CD38+ | 7.1 [3.6 to 9.2]
  %Ki67+ | 0.1 [-0.2 to 0.6]
  %caspase3+ | 0.7 [0.3 to 1.0]
  %Bcl-2- | -0.5 [-0.9 to 0.2]
  %CD57+ | -0.4 [-0.6 to 0.6]

18. Secondary Outcome: Change in Percentage of CD8+ T-cells That Are: naïve (%CD45RA+CCR7+), Central Memory (%CD45RA-CCR7+), Effector Memory (%CD45RA-CCR7-), Effector (%CD45RA+CCR7-), %HLA-DR+CD38+, %CD38+, %Ki67+, %caspase3+, %Bcl-2-, and %CD57+
Description: as for outcome 17
Time Frame: From week 24 to week 48
Population: as for outcome 17
Measure: Median (90% Confidence Interval); unit: % of CD8+ T-cells
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
% of CD8+ T-cells
  naïve (%CD45RA+CCR7+) | 1.1 [-0.8 to 2.2]
  central memory (%CD45RA-CCR7+) | -0.5 [-1.1 to -0.3]
  effector memory (%CD45RA-CCR7-) | -0.1 [-4.0 to 0.5]
  effector (%CD45RA+CCR7-) | 0.4 [-2.1 to 2.1]
  %HLA-DR+CD38+ | 0.1 [-1.5 to 1.3]
  %CD38+ | 4.2 [0.6 to 5.4]
  %Ki67+ | 0.2 [-0.1 to 0.6]
  %caspase3+ | 0.5 [0.2 to 1.1]
  %Bcl-2- | 0 [-0.5 to 0.4]
  %CD57+ | -1.4 [-3.4 to 1.1]

19. Secondary Outcome: Change in Soluble CD14
Description: Change was calculated as the week 24 result (average of the week 22 and week 24 values) minus the baseline result (average of pre-entry and entry values). Soluble CD14 is a marker of gut microbial translocation.
Time Frame: From baseline to week 24
Population: as for outcome 13
Measure: Median (90% Confidence Interval); unit: mcg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
mcg/ml | -0.03 [-0.05 to 0.20]

20. Secondary Outcome: Change in Soluble CD14
Description: Change was calculated as week 36 result minus the week 24 result (average of the week 22 and week 24 values). Soluble CD14 is a marker of gut microbial translocation.
Time Frame: From week 24 to week 36
Population: as for outcome 15
Measure: Median (90% Confidence Interval); unit: mcg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
mcg/ml | -0.17 [-0.40 to 0.05]

21. Secondary Outcome: Change in Soluble CD14
Description: Change was calculated as week 48 result (average of week 46 and week 48) minus the week 24 result (average of the week 22 and week 24 values). Soluble CD14 is a marker of gut microbial translocation.
Time Frame: From week 24 to week 48
Population: as for outcome 17
Measure: Median (90% Confidence Interval); unit: mcg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
mcg/ml | -0.16 [-0.40 to 0.10]

22. Secondary Outcome: Change in High Sensitivity C-reactive Protein (Hs-CRP)
Description: as for outcome 13
Time Frame: From baseline to week 24
Population: as for outcome 13
Measure: Median (90% Confidence Interval); unit: mg/dl
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
mg/dl | 0.01 [-0.02 to 0.07]

23. Secondary Outcome: Change in Interleukin (IL)-6, Monocyte Chemoattractant Protein (MCP)-1, MCP-2, and Plasma CD40 Ligand (CD40L)
Description: as for outcome 13
Time Frame: From baseline to week 24
Population: as for outcome 13
Measure: Median (90% Confidence Interval); unit: pg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
pg/ml
  IL-6 | 0.7 [-0.9 to 1.6]
  MCP-1 | 44.6 [-39.6 to 103.1]
  MCP-2 | -1.4 [-2.4 to 2.2]
  CD40L | -1.8 [-45.6 to 43.1]

24. Secondary Outcome: Change in Intercellular Cell Adhesion Molecule (ICAM)-1, Plasma P-selectin, Soluble TNFRII (sTNFRII), and Matrix Metalloproteinase (MMP)-9
Description: as for outcome 13
Time Frame: From baseline to week 24
Population: as for outcome 13
Measure: Median (90% Confidence Interval); unit: ng/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
ng/ml
  ICAM-1 | -25.7 [-59.3 to 23.5]
  P-selectin | -11.7 [-66.2 to 30.5]
  sTNFRII | 0.18 [0.05 to 0.32]
  MMP-9 | -12.5 [-48.1 to 4.0]

25. Secondary Outcome: Change in D-dimer
Description: as for outcome 13
Time Frame: From baseline to week 24
Population: as for outcome 13
Measure: Median (90% Confidence Interval); unit: mcg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 32
mcg/ml | 0.09 [0.06 to 0.13]

26. Secondary Outcome: Change in Hs-CRP
Description: Change was calculated as week 36 result minus the week 24 result (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 36
Population: as for outcome 15
Measure: Median (90% Confidence Interval); unit: mg/dl
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
mg/dl | -0.01 [-0.04 to 0]

27. Secondary Outcome: Change in IL-6, MCP-1, MCP-2, and Plasma CD40L
Description: Change was calculated as week 36 result minus the week 24 result (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 36
Population: as for outcome 15
Measure: Median (90% Confidence Interval); unit: pg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
pg/ml
  IL-6 | -0.9 [-2.0 to 0.2]
  MCP-1 | -6.9 [-146.5 to 78.6]
  MCP-2 | 0.1 [-3.5 to 3.3]
  CD40L | 0 [-11.3 to 65.5]

28. Secondary Outcome: Change in ICAM-1, Plasma P-selectin, sTNFRII, and MMP-9
Description: Change was calculated as week 36 result minus the week 24 result (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 36
Population: as for outcome 15
Measure: Median (90% Confidence Interval); unit: ng/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
ng/ml
  ICAM-1 | -20.9 [-43.8 to 7.4]
  P-selectin | -13.7 [-49.4 to 67.6]
  sTNFRII | -0.05 [-0.29 to 0.03]
  MMP-9 | 11.3 [-18.7 to 39.8]

29. Secondary Outcome: Change in D-dimer
Description: Change was calculated as week 36 result minus the week 24 result (average of the week 22 and week 24 values).
Time Frame: From week 24 to week 36
Population: as for outcome 15
Measure: Median (90% Confidence Interval); unit: mcg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
mcg/ml | 0.01 [-0.05 to 0.05]

30. Secondary Outcome: Change in Hs-CRP
Description: as for outcome 17
Time Frame: From week 24 to week 48
Population: as for outcome 17
Measure: Median (90% Confidence Interval); unit: mg/dl
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
mg/dl | 0.01 [-0.01 to 0.03]

31. Secondary Outcome: Change in IL-6, MCP-1, MCP-2, and Plasma CD40L
Description: as for outcome 17
Time Frame: From week 24 to week 48
Population: as for outcome 17
Measure: Median (90% Confidence Interval); unit: pg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
pg/ml
  IL-6 | -0.5 [-2.1 to 0.6]
  MCP-1 | 7.7 [-18.5 to 43.2]
  MCP-2 | 0.2 [-2.1 to 1.8]
  CD40L | 32.3 [0 to 66.7]

32. Secondary Outcome: Change in ICAM-1, Plasma P-selectin, sTNFRII, and MMP-9
Description: as for outcome 17
Time Frame: From week 24 to week 48
Population: as for outcome 17
Measure: Median (90% Confidence Interval); unit: ng/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
ng/ml
  ICAM-1 | -32.4 [-46.4 to 6.8]
  P-selectin | -17.3 [-62.1 to 5.2]
  sTNFRII | 0.03 [-0.02 to 0.13]
  MMP-9 | 12.8 [-14.9 to 29.5]

33. Secondary Outcome: Change in D-dimer
Description: as for outcome 17
Time Frame: From week 24 to week 48
Population: as for outcome 17
Measure: Median (90% Confidence Interval); unit: mcg/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
mcg/ml | -0.02 [-0.03 to 0.01]

34. Secondary Outcome: Proportion of Participants With Detectable HIV-1 Viremia as Measured by Single Copy Assay (SCA)
Description: A subject was considered detectable at a specific week if HIV-1 RNA by SCA >=1 copy/ml.
Time Frame: At weeks -1 (pre-entry), 0 (entry), 12, 22, 24, and 36
Population: As-treated: Participants who initiated treatment were included. Through week 24, follow-up while receiving MVC without change in background regimen were included. For week 36, only results obtained while receiving background regimen were included. One subject who had a large rise (blip) in viral load at week 24 was excluded.
Measure: Number; unit: proportion of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 31
proportion of participants
  Week -1 (N=31) | 0.35
  Week 0 (N=31) | 0.32
  Week 12 (N=30) | 0.43
  Week 22 (N=31) | 0.29
  Week 24 (N=29) | 0.48
  Week 36 (N=30) | 0.43

35. Secondary Outcome: Drug Adherence Assessed as Number of Missed Doses Over a 4-day Recall
Description: Self-reported MVC adherence data were based on a four-day (8 expected doses) recall. Based on the wording of the Self Report case report form (CRF), participants reporting that they were currently taking MVC that then failed to complete the record of the number of missed doses were assumed to have no missed doses to report. Missing adherence assessments at a time point of interest were ignored and only those participants completing an adherence assessment at least one time point of interest were included.
Time Frame: At weeks 4, 12, and 24
Population: as for outcome 12
Measure: Median (Full Range); unit: doses missed
Arm/Group | Maraviroc
Number analyzed (Participants) | 33
doses missed
  Week 4 (N=30) | 0 [0 to 8]
  Week 12 (N=28) | 0 [0 to 4]
  Week 24 (N=27) | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: From first dose of MVC until off-study
Description: Grade>=2 signs/symptoms (S/Sx). Diagnoses per ACTG criteria for clinical events & other diseases. Grade>=3 labs. All S/Sx or labs that lead to a change in study treatment. See DAIDS Grading Severity of AEs, V1.0, Dec04, http://rcc.tech-res-intl.com
Arm/Group | Maraviroc
Serious Adverse Events (participants affected / at risk) | 4/34
Other Adverse Events (participants affected / at risk) | 22/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=34)
Bradycardia (Cardiac disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=34)
Abdominal distension (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Pneumonia bacterial (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood albumin abnormal (Investigations) | 2
Blood bilirubin increased (Investigations) | 5
Blood glucose abnormal (Investigations) | 3
Blood glucose increased (Investigations) | 4
Blood sodium decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights